CLINICAL TRIAL: NCT05665933
Title: Acceptance and Commitment Therapy and Test Anxiety in Adolescents
Brief Title: Acceptance and Commitment Therapy and Test Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Artvin Coruh University (Other)
Responsible Party: Principal Investigator, Kubra Tan, Lecturer, Artvin Coruh University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Artvin Coruh U
Record Dates: First submitted 2022-12-07; First posted 2022-12-27 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Therapy, Directly Observed
Keywords: acceptance and commitment therapy; test anxiety; study skills; psychological flexibility
MeSH Terms: conditions — Directly Observed Therapy

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with pretest posttest, experimental and control groups
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THE EFFECT OF ACCEPTANCE AND COMMITMENT THERAPY-BASED PSYCOEDUCATION (Experimental): PSYCHOEDUCATION PROGRAM Total Duration: 6 Weeks Session Duration: 90 min Frequency: 1 day per week Number of People: 30
  Interventions: Behavioral: ACCEPTANCE AND COMMITMENT THERAPY-BASED PSYCOEDUCATION
- THE EFFECT OF ACCEPTANCE AND COMMITMENT THERAPY-BASED PSYCOEDUCATION ON EXAM ANXIETY IN ADOLESCENTS (No Intervention): Similar training will be provided after the study is completed. Number of People: 30

INTERVENTIONS:
Behavioral: ACCEPTANCE AND COMMITMENT THERAPY-BASED PSYCOEDUCATION — Total Duration: 6 Weeks Session Duration: 90 min Frequency: 1 day per week Number of People: 30
  Arms: THE EFFECT OF ACCEPTANCE AND COMMITMENT THERAPY-BASED PSYCOEDUCATION

SUMMARY:
The aim of this study is to evaluate the effect of acceptance and commitment therapy-based psychoeducation on test anxiety, study skills and psychological flexibility on adolescents. test anxiety scale, study skills scale and psychological flexibility scale are data collection tools. The pretest-posttest is a randomized controlled trial. Experimental and control groups were formed. A 6-week psychoeducation will be applied to the experimental group.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of acceptance and commitment therapy-based psychoeducation given to adolescents on test anxiety, study skills and psychological flexibility.The research was designed as a randomized controlled study with pretest, posttest, experimental and control groups aiming to examine the results of Acceptance and Commitment Therapy (ACT) based psychoeducation for test anxiety and study skills. The number of effects of the study was targeted by the randomization method among the adolescents who met the inclusion criteria and accepted the application. In the power analysis, the evaluation of the number of increase is aimed at 0.05 aggression level at the 95% confidence interval, and 52 adolescents, 26 experimental and 26 control groups, to reach 80% power. Randomization methods were used so that individuals could be assigned to the experimental groups with equal chance, similar to the scores they obtained from the laboratory test anxiety periods. 52 adolescents who met the clinical research criteria for randomization were divided into 2 groups using the irregular numbers table, this group was named as the experimental and control groups by drawing lots. The group that came out first in the lottery at this stage was accepted as the experimental group. Psychoeducation is planned to be held between December 2022 and February 2023.

ELIGIBILITY:
Inclusion Criteria:

* Students' willingness to participate in research
* Students being 11th graders
* Getting a score of 50 or more on the test anxiety scale

Exclusion Criteria:

* Any degree of cognitive decline or impairment
* Presence of depressive disorder
* Presence of serious psychiatric disorder
* Being under treatment for a psychiatric condition

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change of Exam Anxiety Scale Total Score | 6 weeks
  Change in test anxiety scale at the end of 6 weeks. The highest score from the test anxiety scale is 80 and the lowest score is 20. A high score defines high anxiety.
Change study skills in adolescents. | 6 weeks
  Change in test study skills scale.A maximum of 165 and a minimum of 55 points are obtained from the study skills scale. A high score defines the ability to study effectively.

SECONDARY OUTCOMES:
Change the level of psychological flexibility | 6 weeks
  Change in test psychological flexibility. A maximum of 196 and a minimum of 28 points are obtained from the psychological flexibility scale. A higher score reflects higher psychological flexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Tan, Study Director — https://www.artvin.edu.tr/kubra-tan
Locations (2):
- Turkey (Türkiye) (2):
  - ArtvinCoruhU, Artvın, Center
  - ArtvinCoruhU, Artvın

IPD SHARING:
Plan to Share IPD: No
The name and results of the study will be shared.